CLINICAL TRIAL: NCT04907773
Title: Evaluation of a Blood Potassium Measurement Device From Capillary Samples
Brief Title: Evaluation of a Blood Potassium Measurement Device From Capillary Samples (ALPHA)
Acronym: ALPHA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CardioRenal (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CR-2021-001
Record Dates: First submitted 2021-05-21; First posted 2021-06-01 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-09

CONDITIONS: Potassium Measurement
Keywords: hemolysis; capillary collection
MeSH Terms: conditions — Hemolysis | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Potassium measurement
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Potassium measurement (Other)
  Interventions: Other: Capillary blood sampling; Other: Venous blood sampling; Other: Arterio-venous blood sampling

INTERVENTIONS:
Other: Capillary blood sampling — Each subject will have one to two capillary blood collections.
Other: Venous blood sampling — Each healthy subject will also have a reference venous blood collection.
Other: Arterio-venous blood sampling — Each hemodialysed subject will also have a reference arterio-venous blood collection.

SUMMARY:
This is an open, prospective, and interventional study investigating the potassium measurement with the CardioRenal device in capillary blood. It will be conducted at one investigational site.

Each subject will have capillary blood collections. Additionally as a reference a venous blood collection will be conducted

DETAILED DESCRIPTION:
Cardiorenal is a company aiming to develop in-vitro diagnostic medical devices to measure the potassium from a single drop of capillary blood to allow an everyday home monitoring of the potassium value like with the diabetes patients who supervise their blood sugar level by measurements with glucose-test stripe from a drop of capillary blood.

A major problem for the blood potassium monitoring at clinical levels is caused by hemolysis leading to the overestimation of potassium level. Hemolysis is the lysis of red blood cells (RBC, erythrocytes) and the release of their contents into plasma. The hemolysis may occur from in vivo or in vitro causes (milking, pressure…). It has also been reported that capillary puncture may induce increased level of hemolysis compared to venous sampling.

CardioRenal aims to limit those factors to guarantee an accurate measurement of potassium concentration in a capillary sample by using a standardized method of capillary pricking.

After clarification the approval the Informed Consent is signed and the inclusion as well as exclusion criteria (incl. demography, concomitant medication and medical history) or vital parameters (weight), are raised.

With 40 healthy subjects capillary and venous blood is taken. Blood is taken from the subject by trained specialist staff. The capillary blood sampling occurs in 400 µl Lithium-Heparin BD vacutainer Microtainers.

* A total of <1mL volume of capillary blood is taken.
* In addition 10 ml blood from the vein of a forearm is taken.

With 30 hemodialysed subjects capillary and venous blood is taken before and/or after dialysis session to extend the potassium concentration range. Blood is taken from the subject by trained specialist staff. The capillary blood sampling occurs in 400 µl Lithium-Heparin BD vacutainer Microtainers.

* A screening based on potassium measurement just before the capillary puncture is performed to test the eligibility of the subject : a 2.5mL blood is taken from the fistula or the central venous catheter.
* A total of <1mL volume of capillary blood is taken.
* In addition 10 ml blood from the fistula or the central venous catheter.

To guarantee a light blood decrease without strong mechanical pressure, the site for capillary puncture are warmed up before the capillary sampling during 2 minutes before puncture.

ELIGIBILITY:
Inclusion Criteria:

* Adults (Age Over 18 yo)
* Healthy volunteers
* Chronic Hemodialysed patients
* Pre-dialysis patient, taken off after the long interdialytic interval (> 2 days)
* AND with a K+ > 5.0 mmol/L just before starting the dialysis session (screening checked on venous or arterio-venous blood sample)
* Post-dialysis, in patients treated with a 2 mmol/l dialysis bath
* AND with a K+ < 3.5 mmol/L at the end of the dialysis session (screening checked on venous or arterio-venous blood sample)

Exclusion Criteria:

* No consent
* Age <18 yo
* Medical history of crisis (epilepsy)
* Known inherited hemolytic anemia
* Autoimmune hemolytic anemia
* Infectious Hemolytic anemia
* Prosthetic Cardiac valves
* Hemolytic uremic syndrome
* Peripheral edema
* Dehydration
* Peripheral Arterial Obstructive Disease (PAOD)
* Raynaud syndrome
* Known evolutive cancers
* Vulnerable patients, patients deprived from liberty and patients with a physical or mental state altered by disease, age or disability which impacts their ability to defend their interests and for which protection measures are taken

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
Correlation between venous whole blood potassium with available point of care device and capillary potassium with CardioRenal device | through study completion, an average of 1 month

SECONDARY OUTCOMES:
Correlation between capillary potassium with available point of care device and capillary potassium with Cardiorenal device | through study completion, an average of 1 month
Correlation between plasma potassium from venous puncture with lab test and capillary potassium with Cardiorenal device | through study completion, an average of 1 month
Correlation between venous whole blood potassium and capillary potassium measurement with available point of care device | through study completion, an average of 1 month
Correlation between plasma potassium from venous puncture with lab test and plasma potassium from venous puncture with Cardiorenal device | through study completion, an average of 1 month

OTHER OUTCOMES:
Correlation from capillary freeHb and capillary potassium | through study completion, an average of 1 month
Degree of haemolysis in capillary blood tests compared to venous blood test | through study completion, an average of 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Damien Gruson, Prof, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques Universitaires Saint-Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No